CLINICAL TRIAL: NCT07055646
Title: Influence of Low Vision Assistive Technology on Mobility Among Visually Impaired Individuals
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/925
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Traditional Assistive Technology
  Interventions: Diagnostic Test: Traditional Assistive Technology
- Digital Assistive Technology
  Interventions: Diagnostic Test: Digital Assistive Technology
- Combined Technology Users
  Interventions: Combination Product: Combined Technology Users

INTERVENTIONS:
Diagnostic Test: Traditional Assistive Technology — Participants in Group 1 utilize traditional, non-digital assistive devices designed to enhance mobility and spatial orientation
  Groups: Traditional Assistive Technology
Diagnostic Test: Digital Assistive Technology — Participants in Group 2 use modern, digital assistive technologies specifically designed to improve navigation, orientation, and real-time decision-making for visually impaired individuals
  Groups: Digital Assistive Technology
Combination Product: Combined Technology Users — Participants in Group 3 use a combination of traditional tools (e.g., cane, magnifiers) alongside modern digital aids (e.g., smart canes, GPS apps). This group is important to examine how integrated usage of both types of technologies
  Groups: Combined Technology Users

SUMMARY:
This study investigates the influence of low vision assistive technology (AT) on the mobility and independence of individuals with visual impairments. The research aims to explore how various low vision devices, such as electronic travel aids, magnifiers, GPS-based navigation tools, and smartphone applications, impact the ability of visually impaired individuals to move safely and confidently within different environments.

DETAILED DESCRIPTION:
The study employs a mixed-methods approach, combining quantitative and qualitative data collection techniques. Quantitatively, surveys and structured questionnaires are administered to a diverse sample of visually impaired participants to assess frequency of AT use, types of devices utilized, and self-reported improvements in mobility. Qualitatively, in-depth interviews and focus group discussions provide deeper insight into user experiences, challenges, and preferences.

ELIGIBILITY:
Inclusion Criteria:

* any age.
* low vision (visual acuity less than 6/18 but equal to or better than 3/60 in the better eye, even with best correction).
* Regular users (minimum 3 months) of at least one type of assistive technology (traditional, digital, or both).
* Able to communicate verbally or in writing (independently or with assistance).
* Willing to provide informed consent and participate in interviews or surveys.

Exclusion Criteria:

* Total blindness (no light perception), as the study focuses on low vision.
* Individuals who have not used any assistive technology for mobility.
* Participants currently enrolled in vision rehabilitation training that could bias the outcomes.
* Those with temporary visual impairment (e.g., post-surgery recovery) rather than permanent low vision.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study employs a mixed-methods approach, combining quantitative and qualitative data collection techniques. Quantitatively, surveys and structured questionnaires are administered to a diverse sample of visually impaired participants to assess frequency of AT use, types of devices utilized, and self-reported improvements in mobility. Qualitatively, in-depth interviews and focus group discussions provide deeper insight into user experiences, challenges, and preferences.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
low vision Orientation and Mobility (O&M) assessment | 12 Months
  A low vision Orientation and Mobility (O&M) assessment evaluates an individual's ability to navigate their environment, considering their vision impairment. These assessments often involve a combination of observation, interviews, and standardized tests to gauge skills in orientation (understanding one's position) and mobility (moving safely). Scoring systems vary, but they generally aim to quantify the level of support needed and track progress over time

CONTACTS AND LOCATIONS:
Locations (1):
- LRBT Tertiary Teaching Eye Hospital (Korangi), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No